CLINICAL TRIAL: NCT04567615
Title: A Phase 2, Randomized, Open-label Study of Relatlimab in Combination With Nivolumab in Participants With Advanced Hepatocellular Carcinoma Who Are Naive to IO Therapy But Progressed on Tyrosine Kinase Inhibitors (RELATIVITY-073)
Brief Title: A Study of Relatlimab in Combination With Nivolumab in Participants With Advanced Liver Cancer Who Have Never Been Treated With Immuno-oncology Therapy After Prior Treatment With Tyrosine Kinase Inhibitors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA224-073; 2018-003151-38 (EudraCT Number); U1111-1218-6499 (Other: UTN Number)
Record Dates: First submitted 2020-09-24; First posted 2020-09-28 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinoma; Hepatoma; Liver Cancer, Adult; Liver Cell Carcinoma; Liver Cell Carcinoma, Adult
Keywords: Hepatocellular Carcinoma; Advanced Hepatocellular Carcinoma; Liver Cancer; Liver Cancer, Adult; Liver Cell Carcinoma; Liver Cell Carcinoma, Adult
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Nivolumab; relatlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm A : Nivolumab (Experimental)
  Interventions: Biological: Nivolumab
- Arm B : Nivolumab + Relatlimab Dose 1 (Experimental)
  Interventions: Biological: Nivolumab; Biological: Relatlimab
- Arm C : Nivolumab + Relatlimab Dose 2 (Experimental)
  Interventions: Biological: Nivolumab; Biological: Relatlimab

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days
  Other Names: OPDIVO, BMS-936558
Biological: Relatlimab — Specified dose on specified days
  Other Names: BMS-986016
  Arms: Arm B : Nivolumab + Relatlimab Dose 1; Arm C : Nivolumab + Relatlimab Dose 2

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of relatlimab in combination with nivolumab in participants with advanced liver cancer who have never been treated with immuno-oncology therapy, after prior treatment with tyrosine kinase inhibitor therapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have a diagnosis of hepatocellular carcinoma (HCC) based on histological confirmation
* Must have advanced/metastatic HCC
* Have to be immunotherapy treatment-naive in the advanced/metastatic setting
* Must have at least one Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 measurable untreated lesion
* Child-Pugh score of 5 or 6
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 for ECOG performance status scale

Key Exclusion Criteria:

* Known fibrolamellar HCC, sarcomatoid HCC, combined hepatocellular cholangiocarcinoma
* Prior organ allograft or allogeneic bone marrow transplantation
* No uncontrolled or significant cardiovascular disease
* No active known autoimmune disease
* Have received one or two lines of tyrosine kinase inhibitor therapies
* Evidence of radiographic progression on or after the last line of tyrosine kinase inhibitor therapy

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2025-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (65):
- Argentina (4):
  - Local Institution - 0010, Ciudad de Buenos Aires, Buenos Aires
  - Local Institution - 0019, Buenos Aires, Distrito Federal
  - Local Institution - 0017, Rosario, Santa Fe Province
  - Local Institution - 0063, San Miguel de Tucumán, Tucumán Province
- Brazil (5):
  - Local Institution - 0025, Belo Horizonte, Minas Gerais
  - Local Institution - 0060, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0016, Barretos, São Paulo
  - Unidade de Pesquisa Clínica do Hospital da Clínicas de Ribeirão Preto-Clinical Oncology, Ribeirão Preto, São Paulo
  - Local Institution - 0015, São Paulo, São Paulo
- Chile (3):
  - Local Institution - 0024, Temuco, Región de la Araucanía
  - Local Institution - 0029, Santiago, Santiago Metropolitan
  - Local Institution - 0018, Santiago, Santiago Metropolitan
- China (6):
  - Local Institution - 0113, Harbin, Heilongjiang
  - Local Institution - 0114, Changsha, Hunan
  - Local Institution - 0118, Xi'an, Shaanxi
  - Local Institution - 0108, Xi'an, Shan3xi
  - Local Institution - 0107, Shanghai, Shanghai Municipality
  - Local Institution - 0117, Hangzhou, Zhejiang
- Czechia (3):
  - Local Institution - 0048, Brno
  - Local Institution - 0047, Hradec Králové
  - Local Institution - 0046, Prague
- France (5):
  - Local Institution - 0069, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Local Institution - 0068, Clichy
  - Local Institution - 0105, Grenoble
  - Local Institution - 0074, Lyon
  - Local Institution - 0067, Pessac
- Hong Kong (2):
  - Local Institution - 0077, Hksar
  - Local Institution - 0079, Shatin
- Japan (6):
  - Local Institution - 0072, Matsuyama, Ehime
  - Local Institution - 0054, Yokohama, Kanagawa
  - Local Institution - 0076, Yokohama, Kanagawa
  - Local Institution - 0045, Ōsaka-sayama, Osaka
  - Local Institution - 0075, Ishikawa
  - Local Institution - 0071, Kyoto
- Mexico (3):
  - Local Institution - 0101, San Luis Potosí City, San Luis Potosí
  - Local Institution - 0100, Cuauhtémoc
  - Local Institution - 0106, Oaxaca City
- Local Institution - 0003, Auckland, New Zealand
- Poland (4):
  - Local Institution - 0013, Krakow, Lesser Poland Voivodeship
  - Local Institution - 0012, Bytom
  - Local Institution - 0009, Mysowice
  - Local Institution - 0039, Warsaw
- Romania (4):
  - Local Institution - 0038, Craiova, Dolj
  - Local Institution - 0037, Bucharest
  - Local Institution - 0036, Cluj-Napoca
  - Local Institution - 0070, Suceava
- Singapore (2):
  - Local Institution - 0001, Singapore, Central Singapore
  - Local Institution - 0004, Singapore
- South Korea (3):
  - Local Institution - 0011, Seoul, Seoul-teukbyeolsi
  - Local Institution - 0020, Seongnam-si
  - Local Institution - 0043, Seoul
- Spain (6):
  - Local Institution - 0050, Donostia / San Sebastian, Gipuzkoa
  - Local Institution - 0066, Barcelona
  - Local Institution - 0073, Córdoba
  - Local Institution - 0051, Madrid
  - Local Institution - 0049, Madrid
  - Local Institution - 0058, Pamplona
- Taiwan (5):
  - Local Institution - 0041, Taichung
  - Local Institution - 0034, Tainan
  - Local Institution - 0031, Taipei
  - Local Institution - 0042, Taipei
  - Local Institution - 0032, Taoyuan District
- Turkey (Türkiye) (3):
  - Local Institution - 0089, Ankara
  - Local Institution - 0090, Edirne
  - Local Institution - 0091, Kadiköy/Istanbul

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 266 Participants Randomized, 264 Treated
Groups:
- Treatment A: Nivolumab 480mg Q4W
- Treatment B: Nivolumab 480mg Q4W + Relatlimab 480mg Q4W
- Treatment C: Nivolumab 480mg Q4W + Relatlimab 960mg Q4W
Period: Randomization
Arm/Group | Treatment A | Treatment B | Treatment C
Started | 128 | 114 | 24
Completed (Completed = received atleast 1 dose of study treatment) | 127 | 113 | 24
Not Completed | 1 | 1 | 0
Not completed — Participant withdrew consent | 1 | 0 | 0
Not completed — Adverse event unrelated to study drug | 0 | 1 | 0
Period: Treatment Period
Arm/Group | Treatment A | Treatment B | Treatment C
Started | 127 | 113 | 24
Completed | 3 | 1 | 0
Not Completed | 124 | 112 | 24
Not completed — Participant Withdrew Consent | 2 | 5 | 1
Not completed — Death | 1 | 2 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Participant No Longer Meets Study Criteria | 0 | 1 | 0
Not completed — Disease Progression | 85 | 63 | 16
Not completed — Study Drug Toxicity | 3 | 10 | 4
Not completed — Adverse Event Unrelated to Study Drug | 11 | 6 | 1
Not completed — Other Reasons | 1 | 2 | 0
Not completed — Still On-going Treatment | 21 | 22 | 2

BASELINE CHARACTERISTICS:
Population: All Randomized Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment A | Treatment B | Treatment C | Total
Number analyzed (Participants) | 128 | 114 | 24 | 266
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.0 (10.4) | 63.3 (11.2) | 68.1 (10.9) | 64.1 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 2 | 46
  Male | 105 | 93 | 22 | 220
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 16 | 0 | 30
  Not Hispanic or Latino | 65 | 47 | 15 | 127
  Unknown or Not Reported | 49 | 51 | 9 | 109
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 61 | 54 | 12 | 127
  Black or African American | 2 | 1 | 0 | 3
  Asian | 28 | 19 | 2 | 49
  American Indian or Alaska Native | 5 | 6 | 0 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Other | 3 | 5 | 0 | 8
  Chinese | 16 | 16 | 4 | 36
  Japanese | 7 | 4 | 3 | 14
  Malay | 0 | 1 | 0 | 1
  Asian Other | 6 | 8 | 2 | 16

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate(ORR) Assessed by BICR
Description: Objective Response Rate (ORR) (as per Recists v1.1) is defined as the percentage of participants whose best overall response (BOR) is either confirmed complete response (CR) or confirmed partial response (PR) based on BICR assessments among all participants in the respective analysis set.
  BOR is defined as the best response, as determined by the BICR, recorded between the date of randomization and the date of first objectively documented progression or death due to any cause or the date of subsequent therapy, whichever occurs first.
  For participants without documented progression or subsequent therapy, all available response designations will contribute to the BOR determination. Confirmation of response is required at least 4 weeks after the initial response.
Time Frame: From randomization to primary completion date (Approximately 29.5 Months)
Population: All Randomized Participants
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 128 | 114 | 24
Percentage | 13.3 [7.9 to 20.4] | 10.5 [5.6 to 17.7] | 12.5 [2.7 to 32.4]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Superiority; Strata adjusted difference in ORR = -2.7, 95% CI 2-sided [-10.7 to 5.3] — Difference in ORR of Treatment B over ORR Treatment A

2. Secondary Outcome: Disease Control Rate Assessed by BICR
Description: Disease Control Rate (DCR) (as per Recists v1.1) is defined as the number of randomized participants who achieve a BOR of confirmed CR, confirmed PR, or stable disease (SD), based on BICR assessments divided by the number of all randomized participants.
Time Frame: From randomization to primary completion date (Approximately 29.5 Months)
Population: All Randomized Participants
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 128 | 114 | 24
Percentage | 44.5 [35.7 to 53.6] | 44.7 [35.4 to 54.3] | 33.3 [15.6 to 55.3]

3. Secondary Outcome: Duration of Response Assessed by BICR
Description: Duration of Response (DOR) (as per Recists v1.1) is defined as the time between the date of first documented response (CR or PR) that is subsequently confirmed, to the date of the first objectively documented tumor progression as determined by the BICR, or death due to any cause, whichever occurs first.
  Participants who die without a reported prior progression will be considered to have an event on the date of their death. Participants who neither progress nor die will be censored on the date of their last evaluable tumor assessment. DOR will be evaluated for responders (confirmed CR or PR) only.
Time Frame: From randomization to primary completion date (Approximately 29.5 Months)
Population: All Confirmed Responders
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 17 | 12 | 3
Months | 5.82 [5.55 to NA] — insufficient number of participants with events to calculate Median. | NA [5.32 to NA] — insufficient number of participants with events to calculate Median and Upper Limit Number. | NA [7.39 to NA] — insufficient number of participants with events to calculate Median and Upper Limit Numbe.

4. Secondary Outcome: Progression Free Survival(PFS) Assessed by BICR
Description: PFS (as per Recists v1.1) is defined as the time between the date of randomization and the date of first documented tumor progression or death due to any cause, whichever occurs first.
  Participants who die without a reported progression will be considered to have progressed on the date of their death.
Time Frame: From randomization to primary completion date (Approximately 29.5 Months)
Population: All Randomized Subjects
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 128 | 114 | 24
Months | 2.00 [1.91 to 3.75] | 2.00 [1.87 to 3.71] | 1.94 [1.74 to 3.71]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Superiority; Cox proportional hazard model = 1.00, 95% CI 2-sided [0.75 to 1.33] — HR of Treatment B over HR Treatment A

5. Secondary Outcome: Objective Response Rate Assessed by Investigator
Description: Objective Response Rate (ORR) (as per Recists v1.1) is defined as the percentage of participants whose best overall response (BOR) is either confirmed complete response (CR) or confirmed partial response (PR) based on investigator assessments among all participants in the respective analysis set.
  BOR is defined as the best response, as determined by the investigator, recorded between the date of randomization and the date of first objectively documented progression or death due to any cause or the date of subsequent therapy, whichever occurs first.
  For participants without documented progression or subsequent therapy, all available response designations will contribute to the BOR determination. Confirmation of response is required at least 4 weeks after the initial response.
Time Frame: From randomization to primary completion date (Approximately 29.5 Months)
Population: All Randomized Participants
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 128 | 114 | 24
Percentage | 14.1 [8.6 to 21.3] | 13.2 [7.6 to 20.8] | 20.8 [7.1 to 42.2]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Superiority; Strata adjusted difference in ORR = -0.9, 95% CI 2-sided [-9.2 to 7.4] — Difference in ORR of Treatment B over ORR Treatment A

6. Secondary Outcome: Disease Control Rate Assessed by Investigator
Description: as for outcome 2
Time Frame: From randomization to primary completion date (Approximately 29.5 Months)
Population: All Randomized Participants
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 128 | 114 | 24
Percentage | 48.4 [39.5 to 57.4] | 50.9 [41.3 to 60.4] | 41.7 [22.1 to 63.4]

7. Secondary Outcome: Duration of Response Assessed by Investigator
Description: Duration of Response (DOR) (as per Recists v1.1) is defined as the time between the date of first documented response (CR or PR) that is subsequently confirmed, to the date of the first objectively documented tumor progression as determined by the investigator, or death due to any cause, whichever occurs first.
  Participants who die without a reported prior progression will be considered to have an event on the date of their death. Participants who neither progress nor die will be censored on the date of their last evaluable tumor assessment. DOR will be evaluated for responders (confirmed CR or PR) only.
Time Frame: From randomization to primary completion date (Approximately 29.5 Months)
Population: All Confirmed Responders
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 18 | 15 | 5
Months | 10.94 [4.63 to NA] — insufficient number of participants with events to calculate Median. to calculate Upper Limit Number. | NA [5.55 to NA] — insufficient number of participants with events to calculate Median. to calculate Median and Upper Limit Number. | 12.42 [3.61 to NA] — insufficient number of participants with events to calculate Median. to calculate Upper Limit Number.

8. Secondary Outcome: Progression Free Survival(PFS) Assessed by Investigator
Description: as for outcome 4
Time Frame: From randomization to primary completion date (Approximately 29.5 Months)
Population: All Randomized Subjects
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 128 | 114 | 24
Months | 3.32 [2.00 to 4.01] | 3.65 [1.97 to 4.30] | 1.94 [1.68 to 3.75]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Superiority; Cox proportional hazard model = 1.00, 95% CI 2-sided [0.75 to 1.33] — HR of Treatment B over HR of Treatment A

9. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time from randomization to the date of death from any cause.
  Overall survival will be censored at the date of randomization for participants who were randomized but had no follow-up.
Time Frame: From randomization to primary completion date (Approximately 29.5 Months)
Population: All Randomized Subjects
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 128 | 114 | 24
Months | 12.68 [9.40 to 18.76] | 12.19 [9.49 to 14.52] | 8.21 [4.76 to 16.92]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Superiority; Cox proportional hazard model = 1.05, 95% CI 2-sided [0.74 to 1.49] — HR of Treatment B over HR of Treatment A

10. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants with an Adverse Event.
  An Adverse Event is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment.
Time Frame: From randomization to primary completion date (Approximately 29.5 Months). Includes events reported between first dose and 30 days after last dose of study therapy.
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 127 | 113 | 24
Participants | 119 | 108 | 22

11. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: Number of participants with Serious Adverse Events
  A serious adverse event is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is an important medical event.
Time Frame: as for outcome 10
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 127 | 113 | 24
Participants | 43 | 46 | 14

12. Secondary Outcome: Number of Participants With Adverse Events Leading to Discontinuation
Description: Number of participants with Adverse Events Leading to Discontinuation
Time Frame: as for outcome 10
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 127 | 113 | 24
Participants | 13 | 14 | 5

13. Secondary Outcome: Death Summary
Description: Number of participants who died.
Time Frame: From randomization to primary completion date (Approximately 29.5 Months)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 127 | 113 | 24
Participants | 67 | 60 | 18

14. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities in Specific Liver Tests
Description: Number of participants with clinical laboratory abnormalities in specific liver tests
Time Frame: as for outcome 10
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 127 | 113 | 24
Participants
  ALT OR AST> 5XULN | 25 | 41 | 6
  ALT OR AST> 10XULN | 7 | 16 | 2
  TOTAL BILIRUBIN > 2XULN: number analyzed (Participants) | 127 | 112 | 24
  TOTAL BILIRUBIN > 2XULN | 17 | 14 | 2
  CONCURRENT ALT OR AST ELEVATION > 3XULN WITH TOTAL BILIRUBIN >2XULN WITHIN 30 DAYS: number analyzed (Participants) | 127 | 112 | 24
  CONCURRENT ALT OR AST ELEVATION > 3XULN WITH TOTAL BILIRUBIN >2XULN WITHIN 30 DAYS | 14 | 10 | 1

15. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities in Thyroid Tests
Description: Number of participants with clinical laboratory abnormalities in thyroid tests
Time Frame: as for outcome 10
Population: All Treated Participants with at least on on-treatment TSH measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 117 | 99 | 18
Participants
  TSH > ULN | 38 | 42 | 2
  TSH > ULN WITH TSH ≤ ULN AT BASELINE | 14 | 18 | 1
  TSH <LLN WITH TSH ≥ LLN AT BASELINE | 16 | 26 | 2

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events: (From first dose to last dose to primary completion date) : Approximately 29.5 months All-Cause mortality (From randomization to primary completion date): Approximately 29.5 months
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Arm/Group | Treatment A | Treatment B | Treatment C
All-Cause Mortality (participants affected / at risk) | 68/128 | 60/114 | 18/24
Serious Adverse Events (participants affected / at risk) | 65/127 | 65/113 | 20/24
Other Adverse Events (participants affected / at risk) | 104/127 | 102/113 | 22/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=127) | Treatment B (N=113) | Treatment C (N=24)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 2 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Heart valve incompetence (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0
Myocarditis (Cardiac disorders) | 0 | 1 | 2
Myopericarditis (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 1 | 0
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 0 | 1 | 0
Glucocorticoid deficiency (Endocrine disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0
Ascites (Gastrointestinal disorders) | 3 | 3 | 1
Colitis (Gastrointestinal disorders) | 0 | 2 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0
Colitis microscopic (Gastrointestinal disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 2 | 1 | 0
Haemoperitoneum (Gastrointestinal disorders) | 1 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 3 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Adverse event (General disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 2 | 1 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 2 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Hepatobiliary disease (Hepatobiliary disorders) | 1 | 0 | 0
Hepatorenal failure (Hepatobiliary disorders) | 2 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 2 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0
Liver injury (Hepatobiliary disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Abdominal wall abscess (Infections and infestations) | 1 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 1 | 0
COVID-19 (Infections and infestations) | 3 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Groin abscess (Infections and infestations) | 0 | 1 | 0
Liver abscess (Infections and infestations) | 0 | 1 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 5 | 3 | 1
Pneumonia aspiration (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 2 | 0 | 1
Spontaneous bacterial peritonitis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
General physical condition abnormal (Investigations) | 3 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 1
Troponin T increased (Investigations) | 0 | 1 | 0
Troponin increased (Investigations) | 0 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Necrotising myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Liver carcinoma ruptured (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 29 | 24 | 6
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0
Immune-mediated myasthenia gravis (Nervous system disorders) | 0 | 1 | 0
Monoplegia (Nervous system disorders) | 1 | 0 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 4 | 1
Azotaemia (Renal and urinary disorders) | 0 | 1 | 0
Glomerulonephritis (Renal and urinary disorders) | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0
Shock haemorrhagic (Vascular disorders) | 2 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=127) | Treatment B (N=113) | Treatment C (N=24)
Anaemia (Blood and lymphatic system disorders) | 21 | 16 | 6
Leukopenia (Blood and lymphatic system disorders) | 2 | 4 | 2
Lymphopenia (Blood and lymphatic system disorders) | 8 | 3 | 2
Neutropenia (Blood and lymphatic system disorders) | 3 | 7 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 9 | 2
Hyperthyroidism (Endocrine disorders) | 1 | 9 | 1
Hypothyroidism (Endocrine disorders) | 5 | 15 | 1
Abdominal pain (Gastrointestinal disorders) | 10 | 16 | 2
Abdominal pain upper (Gastrointestinal disorders) | 6 | 5 | 3
Ascites (Gastrointestinal disorders) | 6 | 11 | 4
Constipation (Gastrointestinal disorders) | 12 | 12 | 1
Diarrhoea (Gastrointestinal disorders) | 11 | 20 | 6
Dry mouth (Gastrointestinal disorders) | 2 | 6 | 0
Nausea (Gastrointestinal disorders) | 6 | 17 | 2
Vomiting (Gastrointestinal disorders) | 4 | 7 | 0
Asthenia (General disorders) | 16 | 9 | 7
Fatigue (General disorders) | 16 | 16 | 3
Oedema peripheral (General disorders) | 17 | 20 | 2
Pyrexia (General disorders) | 8 | 9 | 2
Hypertransaminasaemia (Hepatobiliary disorders) | 2 | 6 | 1
COVID-19 (Infections and infestations) | 7 | 14 | 3
Respiratory tract infection (Infections and infestations) | 0 | 1 | 2
Urinary tract infection (Infections and infestations) | 4 | 8 | 2
Alanine aminotransferase increased (Investigations) | 21 | 27 | 3
Amylase increased (Investigations) | 5 | 13 | 2
Aspartate aminotransferase increased (Investigations) | 33 | 33 | 3
Blood alkaline phosphatase increased (Investigations) | 8 | 6 | 0
Blood bilirubin increased (Investigations) | 14 | 18 | 3
Blood creatinine increased (Investigations) | 9 | 10 | 3
Lipase increased (Investigations) | 8 | 12 | 3
Platelet count decreased (Investigations) | 4 | 10 | 1
Troponin increased (Investigations) | 2 | 6 | 1
Decreased appetite (Metabolism and nutrition disorders) | 10 | 15 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 8 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 8 | 4 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 | 8 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 8 | 9 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 11 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 13 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 8 | 1
Headache (Nervous system disorders) | 7 | 5 | 0
Insomnia (Psychiatric disorders) | 2 | 5 | 3
Proteinuria (Renal and urinary disorders) | 6 | 8 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 8 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 24 | 16 | 4
Rash (Skin and subcutaneous tissue disorders) | 8 | 12 | 4
Hypertension (Vascular disorders) | 5 | 6 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-26): https://cdn.clinicaltrials.gov/large-docs/15/NCT04567615/Prot_SAP_000.pdf